CLINICAL TRIAL: NCT06321588
Title: Autoimmune Dementia: Predictors of Neuronal Synaptic Antibodies in Patients With New-ONset Cognitive Impairment and Their Relevance in Non-encephalitic formS: The ADONIS Study
Brief Title: Autoimmune Dementia: Predictors of Neuronal Synaptic Antibodies in Patients With New-ONset Cognitive Impairment
Acronym: ADONIS
Status: Recruiting | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: GR-2021-12373134
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort: patients with a diagnosis of new-onset neurocognitive disorders (major and minor) with onset within the previous 24 months
- prospective cohort: patients with a diagnosis of new-onset neurocognitive disorders (major and minor) with onset within the previous 24 months

SUMMARY:
The goal of this observational study is to investigate the frequency and the possible pathogenic role of neuronal synaptic antibodies (NSAb) in patients with cognitive impairment (CI). The main questions it aims to answer are:

1. the frequency and associated features of NSAb in patients with CI and the usefulness of a clinical score in improving autoimmune dementia (AID) diagnosis;
2. the clinical significance of NSAb in patients with CI not fulfilling the autoimmune encephalitis (AE) criteria and serum NSAb (NSAb-pos-CI);
3. the impact of blood-brain-barrier (BBB) dysfunction on their pathogenicity.

DETAILED DESCRIPTION:
AE can mimic dementia and, contrarily to neurodegenerative dementia syndromes, affected patients can improve with timely immunotherapies. Consensus-based diagnostic criteria for AE help to select patients for antibody testing. However, encephalitis signs can be absent, particularly in the elderly, and AE can present with slowly progressing CI mimicking classical neurodegenerative diseases, misleading the diagnostic process. Data on the prevalence of NSAb and AE in unselected patients with CI are sparse and mostly affected by retrospective design, small cohorts, and antibody assay shortcomings. There is an urgent need to define the frequency of NSAb and AE in CI patients and elucidate the associated clinical, laboratory and imaging features. Filling these gaps is the first aim of this project. This will allow the early identification and the best management of patients with AID. On the other hand, a proportion of CI patients have NSAb and do not fit the AE criteria (NSAb-pos-CI).

These NSAb are often in the serum, and not in the Cerebrospinal Fluid (CSF), or belong to the Immunoglobulin A/M (Ig A/M) subclasses, as opposite to the AE-associated Immunoglobulin G (IgG) subclass, thus triggering questions about their clinical and therapeutic implications. As NSAb can be found at low titers in the serum of healthy controls, a hypothesis explaining their pathogenicity relies on dysfunctions of the BBB, in a context of indolent inflammation, that might allow the antibodies to reach the Central Nervous System (CNS). Alternatively, NSAb may not be directly pathogenic and could even be secondary to an ongoing neurodegenerative process. However, even in this context, known and unknown NSAb, could still contribute to the clinical phenotype, modulating the disease progression or the presence of additional clinical features (i.e. psychiatric symptoms). Understanding if these serum NSAb, along with other factors such as inflammation and BBB alterations, have a role in modifying the disease trajectory, i.e. accelerating the neurodegeneration and CI progression, is the other main goal. This project will represent a chance to clarify the role of NSAb in NSAb-pos-CI and potentially help to identify a subgroup of patients with specific phenotypes, who could benefit from immunotherapies. The identification of such patients will allow their best clinical management.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* adult (aged between 40 and 90 years)
* patients with a diagnosis of new-onset neurocognitive disorders (major and minor), as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, with onset within the previous 24 months

Exclusion Criteria:

- presence of a history of seizures within 4 weeks from onset.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of new-onset neurocognitive disorders (major and minor)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
frequency of antibodies against neuronal antigens | at baseline
  NSAb frequency will be calculated by dividing the number of patients with NSAb with the total number of patients
frequency of antibodies against neuronal antigens | 12 months (54 weeks)
  NSAb frequency will be calculated by dividing the number of patients with NSAb with the total number of patients
creation of a score that predicts the presence of NSAb | 24 months (108 weeks)
  Based on logistic regression models including the clinical, imaging and biomarkers data. The minimum and maximum score is to be defined on the bases of the analyses of the clinical data at 24 months milestone.An higher score is expected to be associated with the antibody presence.

SECONDARY OUTCOMES:
changes of neurodegeneration biomarkers | at baseline
  comparison of blood biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The blood biomarkers are: phosphorylated tau protein 181 (p-tau 181) (pg/mL), Neurofilament Light chain (NfL) (pg/mL), Glial Fibrillary Acidic Protein (GFAP) (pg/mL).
changes of neurodegeneration biomarkers | 1 year (54 weeks)
  comparison of blood biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The blood biomarkers are: phosphorylated tau protein 181 (p-tau 181) (pg/mL), Neurofilament Light chain (NfL) (pg/mL), Glial Fibrillary Acidic Protein (GFAP) (pg/mL).
changes of neuroanatomy | at baseline
  comparison of Brain MRI from baseline to one year follow up in seropositive versus seronegative patients
changes of neuroanatomy | 1 year (54 weeks)
  comparison of Brain MRI from baseline to one year follow up in seropositive versus seronegative patients
changes of inflammatory biomarkers | at baseline
  comparison of inflammatory biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The inflammatory biomarkers are: Interferon alpha (IFN alpha) (pg/mL), Interferon gamma (IFN gamma) (pg/mL), Interleukin-1 beta (IL-1 beta) (pg/mL), Interleukin-2 (IL-2) (pg/mL), Interleukin-4 (IL-4) (pg/mL), Interleukin-5 (IL-5) (pg/mL), Interleukin-6 (IL-6) (pg/mL), Interleukin-8 (IL-8) (pg/mL), Interleukin-17A (IL-17A) (pg/mL), Tumor necrosis factor alpha (TNF alpha) (pg/mL), Interferon gamma-induced protein 10 (IP-10) known as C-X-C motif chemokine 10(CXCL10) (pg/mL), Monocyte chemoattractant protein-1 (MCP-1) known as C-C motif chemokine ligand 2 (CCL2) (pg/mL).
changes of inflammatory biomarkers | 1 year (54 weeks)
  comparison of inflammatory biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The inflammatory biomarkers are: Interferon alpha (IFN alpha) (pg/mL), Interferon gamma (IFN gamma) (pg/mL), Interleukin-1 beta (IL-1 beta) (pg/mL), Interleukin-2 (IL-2) (pg/mL), Interleukin-4 (IL-4) (pg/mL), Interleukin-5 (IL-5) (pg/mL), Interleukin-6 (IL-6) (pg/mL), Interleukin-8 (IL-8) (pg/mL), Interleukin-17A (IL-17A) (pg/mL), Tumor necrosis factor alpha (TNF alpha) (pg/mL), Interferon gamma-induced protein 10 (IP-10) known as C-X-C motif chemokine 10(CXCL10) (pg/mL), Monocyte chemoattractant protein-1 (MCP-1) known as C-C motif chemokine ligand 2 (CCL2) (pg/mL).
changes of brain blood barrier biomarkers | at baseline
  comparison of brain blood barrier biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The biomarkers are: S100 calcium-binding protein B (S-100b) (pg/mL), Glial Fibrillary Acidic Protein (GFAP) (pg/mL).
changes of brain blood barrier biomarkers | 1 year (54 weeks)
  comparison of brain blood barrier biomarkers from baseline to one year follow up in seropositive versus seronegative patients. The biomarkers are: S100 calcium-binding protein B (S-100b) (pg/mL), Glial Fibrillary Acidic Protein (GFAP) (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pia Giannoccaro, Dr., Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (3):
- Italy (3):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Bologna
  - Istituto Auxologico Italiano IRCCS, Milan, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bartels F, Stronisch T, Farmer K, Rentzsch K, Kiecker F, Finke C. Neuronal autoantibodies associated with cognitive impairment in melanoma patients. Ann Oncol. 2019 May 1;30(5):823-829. doi: 10.1093/annonc/mdz083. PMID 30840061
- [Result] Brunkhorst R, Pfeilschifter W, Foerch C. Astroglial proteins as diagnostic markers of acute intracerebral hemorrhage-pathophysiological background and clinical findings. Transl Stroke Res. 2010 Dec;1(4):246-51. doi: 10.1007/s12975-010-0040-6. Epub 2010 Aug 28. PMID 24323552
- [Result] Castillo-Gomez E, Oliveira B, Tapken D, Bertrand S, Klein-Schmidt C, Pan H, Zafeiriou P, Steiner J, Jurek B, Trippe R, Pruss H, Zimmermann WH, Bertrand D, Ehrenreich H, Hollmann M. All naturally occurring autoantibodies against the NMDA receptor subunit NR1 have pathogenic potential irrespective of epitope and immunoglobulin class. Mol Psychiatry. 2017 Dec;22(12):1776-1784. doi: 10.1038/mp.2016.125. Epub 2016 Aug 9. PMID 27502473
- [Result] Constantinescu R, Krysl D, Bergquist F, Andren K, Malmestrom C, Asztely F, Axelsson M, Menachem EB, Blennow K, Rosengren L, Zetterberg H. Cerebrospinal fluid markers of neuronal and glial cell damage to monitor disease activity and predict long-term outcome in patients with autoimmune encephalitis. Eur J Neurol. 2016 Apr;23(4):796-806. doi: 10.1111/ene.12942. Epub 2016 Jan 29. PMID 26822123
- [Result] Dubey D, Kothapalli N, McKeon A, Flanagan EP, Lennon VA, Klein CJ, Britton JW, So E, Boeve BF, Tillema JM, Sadjadi R, Pittock SJ. Predictors of neural-specific autoantibodies and immunotherapy response in patients with cognitive dysfunction. J Neuroimmunol. 2018 Oct 15;323:62-72. doi: 10.1016/j.jneuroim.2018.07.009. Epub 2018 Jul 25. PMID 30196836
- [Result] Dubois B, Villain N, Frisoni GB, Rabinovici GD, Sabbagh M, Cappa S, Bejanin A, Bombois S, Epelbaum S, Teichmann M, Habert MO, Nordberg A, Blennow K, Galasko D, Stern Y, Rowe CC, Salloway S, Schneider LS, Cummings JL, Feldman HH. Clinical diagnosis of Alzheimer's disease: recommendations of the International Working Group. Lancet Neurol. 2021 Jun;20(6):484-496. doi: 10.1016/S1474-4422(21)00066-1. Epub 2021 Apr 29. PMID 33933186
- [Result] Flanagan EP, McKeon A, Lennon VA, Boeve BF, Trenerry MR, Tan KM, Drubach DA, Josephs KA, Britton JW, Mandrekar JN, Lowe V, Parisi JE, Pittock SJ. Autoimmune dementia: clinical course and predictors of immunotherapy response. Mayo Clin Proc. 2010 Oct;85(10):881-97. doi: 10.4065/mcp.2010.0326. PMID 20884824
- [Result] Giannoccaro MP, Cossins J, Sorland K, Fluge O, Vincent A. Searching for Serum Antibodies to Neuronal Proteins in Patients With Myalgic Encephalopathy/Chronic Fatigue Syndrome. Clin Ther. 2019 May;41(5):836-847. doi: 10.1016/j.clinthera.2019.04.001. Epub 2019 May 1. PMID 31053295
- [Result] Gibson LL, McKeever A, Cullen AE, Nicholson TR, Aarsland D, Zandi MS, Pollak TA. Neuronal surface autoantibodies in dementia: a systematic review and meta-analysis. J Neurol. 2021 Aug;268(8):2769-2779. doi: 10.1007/s00415-020-09825-0. Epub 2020 Apr 18. PMID 32306172
- [Result] Pollak TA, Vincent A, Iyegbe C, Coutinho E, Jacobson L, Rujescu D, Stone J, Jezequel J, Rogemond V, Jamain S, Groc L, David A, Egerton A, Kahn RS, Honnorat J, Dazzan P, Leboyer M, McGuire P. Relationship Between Serum NMDA Receptor Antibodies and Response to Antipsychotic Treatment in First-Episode Psychosis. Biol Psychiatry. 2021 Jul 1;90(1):9-15. doi: 10.1016/j.biopsych.2020.11.014. Epub 2020 Nov 24. PMID 33536130
- [Result] Wagner J, Witt JA, Helmstaedter C, Malter MP, Weber B, Elger CE. Automated volumetry of the mesiotemporal structures in antibody-associated limbic encephalitis. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):735-42. doi: 10.1136/jnnp-2014-307875. Epub 2014 Sep 2. PMID 25185210
- [Result] Yeshokumar AK, Gordon-Lipkin E, Arenivas A, Cohen J, Venkatesan A, Saylor D, Probasco JC. Neurobehavioral outcomes in autoimmune encephalitis. J Neuroimmunol. 2017 Nov 15;312:8-14. doi: 10.1016/j.jneuroim.2017.08.010. Epub 2017 Aug 31. PMID 28889962